CLINICAL TRIAL: NCT02351700
Title: Randomized, Double-Blind, Placebo-Controlled Trial Comparing Opioid-Sparing and Opioid-Containing Analgesia Regimens Following Trans-sphenoidal Surgery for Pituitary Tumors
Brief Title: Analgesia Regimens Following Trans-sphenoidal Surgery for Pituitary Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14BN090
Record Dates: First submitted 2015-01-14; First posted 2015-01-30 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2019-11

CONDITIONS: Pituitary Tumor; Pain
MeSH Terms: conditions — Pituitary Neoplasms; Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Caldolor (ibuprofen) (Active Comparator): Intravenous (IV) Caldolor (ibuprofen) (800mg every 8 hours) initiated during surgery and oral acetaminophen 1000mg every 6 hours initiated post-operatively and continued for the duration of the hospital stay (an expected average stay of 2 days) or 48 hours, whichever comes first. Breakthrough pain will be treated with rescue narcotics (IV morphine 2-4mg every 2 hours and oral oxycodone 5-15mg every 4 hours immediately post-operatively through discharge, an expected average stay of 2 days). Hydromorphone (IV 0.5-2mg every 2 hours and oral 2-4mg every 4 hours) will be used in patients with morphine or oxycodone allergy or intolerance.
  Interventions: Drug: IV Caldolor
- standard treatment group (Placebo Comparator): IV placebo will be initiated during surgery and oral acetaminophen 1000mg every 6 hours will be initiated post-operatively and continued for the duration of the hospital stay (an expected average stay of 2 days) or 48 hours, whichever comes first. Breakthrough pain will be treated with rescue narcotics (IV morphine 2-4mg every 2 hours and oral oxycodone 5-15mg every 4 hours immediately post-operatively through discharge, an expected average stay of 2 days). Hydromorphone (IV 0.5-2mg every 2 hours and oral 2-4mg every 4 hours) will be used in patients with morphine or oxycodone allergy or intolerance.
  Interventions: Drug: IV Placebo

INTERVENTIONS:
Drug: IV Caldolor — IV Caldolor (IV ibuprofen) intraoperatively and postoperatively
  Other Names: IV ibuprofen; Opioid Sparing group
  Arms: IV Caldolor (ibuprofen)
Drug: IV Placebo — IV Placebo intraoperatively and postoperatively
  Other Names: Standard treatment group
  Arms: standard treatment group

SUMMARY:
A randomized, double-blind, placebo-controlled intervention trial involving 100 treated subjects undergoing endonasal trans-sphenoidal (ENTS) resection of pituitary lesion. Subjects will be randomized into two groups: 50 treated in the opioid-sparing arm and 50 treated in the standard post-operative medication arm.

DETAILED DESCRIPTION:
Post-operative pain control is a common concern patients have when they consider undergoing a surgical procedure. Although effective for treating acute pain, opioid analgesics are also associated with dose-dependent adverse effects, including constipation, nausea and vomiting, altered mental status, and respiratory depression, all of which have been shown to increase patient length of stay. The use of non-opioid analgesics with different mechanisms of actions for acute pain control via a multi-modal approach is efficacious in reducing opioid consumption, decreasing the incidence of adverse effects, improving patient satisfaction and recovery time, and decreasing hospital costs.Certain minimally invasive procedures may afford many patients the opportunity to achieve adequate post-operative pain control with minimal to no requirement of opioid analgesics, thereby sparing the patient known adverse effects that can increase length of stay and costs. The ENTS approach for resection of pituitary tumors is the standard surgical procedure for these lesions, and is associated with pain that is more easily managed post-operatively, making it an ideal procedure for an opioid-sparing post-operative pain regimen. Anecdotally, the investigators note that in the investigator's post-operative pituitary patient population that post-operative pain can frequently be adequately managed with scheduled non-opioid analgesics, often without requiring breakthrough opioid doses. Another safe and effective non-opioid analgesic that is widely used in multi-modal pain management for moderate pain is IV Caldolor (ibuprofen). After literature review, the investigators were unable to find a study that had attempted to use an opioid-sparing analgesic regimen for post-operative pain control following ENTS approach for resection of pituitary tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing ENTS surgery for resection of pituitary tumor.
* Adults >18 years and <80 years of age.
* English speaking and literate or able to understand the use of a pain scale.
* Body Mass Index >19 and <40 kg/m2

Exclusion Criteria:

* Renal failure (acute or chronic) or creatinine >2.0
* Allergy or intolerance to acetaminophen, ibuprofen, or opioids
* Pre-operative opioid tolerance, dependence, or abuse
* Anaphylaxis to opioids
* History of peptic ulcer disease or recent gastrointestinal bleed requiring surgery
* Cirrhosis, hepatitis, liver transplant, or liver function studies out of normal range, defined as aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/bilirubin> 3x upper limit of normal range
* Subject unwilling or unable to sign informed consent for the study
* Pregnancy
* Incarcerated patients

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Little, MD, Principal Investigator — Barrow Neurosurgical Associates physician with SJHMC privileges
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Pizzi LT, Toner R, Foley K, Thomson E, Chow W, Kim M, Couto J, Royo M, Viscusi E. Relationship between potential opioid-related adverse effects and hospital length of stay in patients receiving opioids after orthopedic surgery. Pharmacotherapy. 2012 Jun;32(6):502-14. doi: 10.1002/j.1875-9114.2012.01101.x. Epub 2012 May 8. PMID 22570188
- [Background] Husted H. Fast-track hip and knee arthroplasty: clinical and organizational aspects. Acta Orthop Suppl. 2012 Oct;83(346):1-39. doi: 10.3109/17453674.2012.700593. PMID 23205862
- [Background] Costantini R, Affaitati G, Fabrizio A, Giamberardino MA. Controlling pain in the post-operative setting. Int J Clin Pharmacol Ther. 2011 Feb;49(2):116-27. doi: 10.5414/cp201401. PMID 21255528
- [Background] Badie B, Nguyen P, Preston JK. Endoscopic-guided direct endonasal approach for pituitary surgery. Surg Neurol. 2000 Feb;53(2):168-72; discussion 172-3. doi: 10.1016/s0090-3019(99)00195-0. PMID 10713196
- [Background] Dahl V, Dybvik T, Steen T, Aune AK, Rosenlund EK, Raeder JC. Ibuprofen vs. acetaminophen vs. ibuprofen and acetaminophen after arthroscopically assisted anterior cruciate ligament reconstruction. Eur J Anaesthesiol. 2004 Jun;21(6):471-5. doi: 10.1017/s026502150400609x. PMID 15248627
- [Background] Southworth S, Peters J, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen 400 and 800 mg every 6 hours in the management of postoperative pain. Clin Ther. 2009 Sep;31(9):1922-35. doi: 10.1016/j.clinthera.2009.08.026. PMID 19843482
- [Background] Singla N, Rock A, Pavliv L. A multi-center, randomized, double-blind placebo-controlled trial of intravenous-ibuprofen (IV-ibuprofen) for treatment of pain in post-operative orthopedic adult patients. Pain Med. 2010 Aug;11(8):1284-93. doi: 10.1111/j.1526-4637.2010.00896.x. Epub 2010 Jun 30. PMID 20609131
- [Background] Kroll PB, Meadows L, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen (i.v.-ibuprofen) in the management of postoperative pain following abdominal hysterectomy. Pain Pract. 2011 Jan-Feb;11(1):23-32. doi: 10.1111/j.1533-2500.2010.00402.x. PMID 20642488
- [Background] Chung KC, Barlev A, Braun AH, Qian Y, Zagari M. Assessing analgesic use in patients with advanced cancer: development of a new scale--the Analgesic Quantification Algorithm. Pain Med. 2014 Feb;15(2):225-32. doi: 10.1111/pme.12299. Epub 2014 Jan 8. PMID 24400921
- [Result] Shepherd DM, Jahnke H, White WL, Little AS. Randomized, double-blinded, placebo-controlled trial comparing two multimodal opioid-minimizing pain management regimens following transsphenoidal surgery. J Neurosurg. 2018 Feb;128(2):444-451. doi: 10.3171/2016.10.JNS161355. Epub 2017 Mar 3. PMID 28298041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients undergoing endonasal transsphenoidal surgery for pituitary adenoma. Potential patients were identified in the Pituitary Clinic at Barrow Neurological Institute.
Pre-assignment Details: Randomized 1:1 ratio with blinded treatment assignment. Used a computer-generated list from random.org.
Groups:
- Opioid-sparing Group: Intravenous (IV) Caldolor (ibuprofen) (800mg every 8 hours) initiated during surgery and oral acetaminophen 1000mg every 6 hours initiated post-operatively and continued for the duration of the hospital stay (an expected average stay of 2 days) or 48 hours, whichever comes first. Breakthrough pain will be treated with rescue narcotics (IV morphine 2-4mg every 2 hours and oral oxycodone 5-15mg every 4 hours immediately post-operatively through discharge, an expected average stay of 2 days). Hydromorphone (IV 0.5-2mg every 2 hours and oral 2-4mg every 4 hours) will be used in patients with morphine or oxycodone allergy or intolerance.
  IV Caldolor (IV Ibuprofen): Compare addition of IV Caldolor (IV ibuprofen) intraoperatively and postoperatively against IV ibuprofen placebo added intraoperatively and postoperatively.
- Standard Treatment Group: IV Caldolor placebo will be initiated during surgery and oral acetaminophen 1000mg every 6 hours will be initiated post-operatively and continued for the duration of the hospital stay (an expected average stay of 2 days) or 48 hours, whichever comes first. Breakthrough pain will be treated with rescue narcotics (IV morphine 2-4mg every 2 hours and oral oxycodone 5-15mg every 4 hours immediately post-operatively through discharge, an expected average stay of 2 days). Hydromorphone (IV 0.5-2mg every 2 hours and oral 2-4mg every 4 hours) will be used in patients with morphine or oxycodone allergy or intolerance.
  IV Ibuprofen placebo: Compare addition of IV ibuprofen placebo intraoperatively and postoperatively against IV Caldolor (IV ibuprofen) added intraoperatively and postoperatively.
Period: Overall Study
Arm/Group | Opioid-sparing Group | Standard Treatment Group
Started | 28 | 34
Completed | 28 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients age >18 years and <80 years undergoing endonasal transsphenoidal surgery for pituitary adenoma.
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid-sparing Group | Standard Treatment Group | Total
Number analyzed (Participants) | 28 | 34 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 29 | 43
  >=65 years | 14 | 5 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 30 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 34 | 62

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Mean Pain Scores Between Two Arms (Measured Every 4 Hours Over 48 Hour)
Description: Comparison of pain scores between two arms using Visual Analog Scale (VAS) for Pain. Units of measure are 0=No Pain, 1=Annoying, 2=Mild Pain, 3=Troublesome, 4=Nagging Pain, Uncomfortable, 5=Distressing, 6=Miserable, 7=Horrible, 8=Intense, Dreadful, 9=Unbearable, 10=Worst Possible Pain. Higher values represent a worse outcome. There are no subscales.
Time Frame: mean pain score over 48 hours
Population: All participants enrolled with the intent to treat.
Measure: Mean (Standard Deviation); unit: 0-10 units on a scale
Arm/Group | Opioid-sparing Group | Standard Treatment Group
Number analyzed (Participants) | 28 | 34
0-10 units on a scale | 1.7 (2.2) | 2.8 (3.0)

2. Secondary Outcome: Breakthrough Narcotic Requirement
Description: Rescue narcotic in both groups will be recorded and compared using a standard equianalgesic oral morphine equivalent (OME) calculation
Time Frame: until discharge from hospital, an expected stay of 2 days
Population: All participants enrolled with the intent to treat.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Opioid-sparing Group | Standard Treatment Group
Number analyzed (Participants) | 28 | 34
mg | 26.3 (28.7) | 62.5 (63.8)

3. Secondary Outcome: Other Adverse Events
Description: Epistaxis, potentially related to IV ibuprofen, will be compared between two groups
Time Frame: until discharge from hospital, an expected stay of 2 days
Measure: Number; unit: participants
Groups:
- Opioid Sparing Group: IV Caldolor (ibuprofen) 800 mg every 8 hours initiated during surgery and oral acetaminophen 1000 mg every 6 hours plus rescue opiates as needed
- Standard Treatment Group: IV placebo every 8 hours initiated during surgery and oral acetaminophen 1000 mg every 6 hours plus rescue opiates as needed
Arm/Group | Opioid Sparing Group | Standard Treatment Group
Number analyzed (Participants) | 28 | 34
participants | 0 | 2

4. Other Pre Specified Outcome: Total Cost of Hospital Charges Compared Between Two Arms
Description: Total hospital costs for patients in IV ibuprofen arm compared to IV placebo arm
Time Frame: until discharge from hospital, an expected stay of 2 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: The Number of Participants Who Have a Bowel Movement During Hospitalization in Both Groups
Description: patients with one or more bowel movement(s) in the first 48 hours after surgery
Time Frame: until discharge from hospital, an expected stay of 2 days
Population: all patients enrolled with intent to treat
Measure: Number; unit: participants
Arm/Group | Opioid-sparing Group | Standard Treatment Group
Number analyzed (Participants) | 28 | 34
participants | 9 | 12

6. Other Pre Specified Outcome: Length of Stay in Hospital Compared Between Two Arms
Description: Length of hospital stay from time of surgery to time of discharge.
Time Frame: until discharge from hospital, an expected stay of 2 days
Population: all participants enrolled with the intent to treat
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Opioid-sparing Group | Standard Treatment Group
Number analyzed (Participants) | 28 | 34
hours | 71.3 (47.5) | 51.7 (30.3)

7. Other Pre Specified Outcome: Total Number of Doses of Any Anti-emetic Required Post-operatively in Both Groups
Description: Use of antiemetics in first 48 hours after surgery
Time Frame: until discharge from hospital, an expected stay of 2 days
Population: all participants enrolled with the intent to treat
Measure: Mean (Standard Deviation); unit: dose
Arm/Group | Opioid-sparing Group | Standard Treatment Group
Number analyzed (Participants) | 28 | 34
dose | 9.8 (9.1) | 10.1 (6.6)

ADVERSE EVENTS:
Time Frame: surgery date until hospital discharge (average of 2 days)
Groups:
- Opioid-sparing Group: Intravenous (IV) Caldolor (ibuprofen) (800mg every 8 hours) initiated during surgery and oral acetaminophen 1000mg every 6 hours initiated post-operatively and continued for the duration of the hospital stay (an expected average stay of 2 days) or 48 hours, whichever comes first. Breakthrough pain will be treated with rescue narcotics (IV morphine 2-4 mg every 2 hours and oral oxycodone 5-15mg every 4 hours immediately post-operatively through discharge, an expected average stay of 2 days). Hydromorphone (IV 0.5-2 mg every 2 hours and oral 2-4 mg every 4 hours) will be used in patients with morphine or oxycodone allergy or intolerance.
  IV Caldolor (Ibuprofen): Compare addition of IV Caldolor (ibuprofen) intraoperatively and postoperatively against IV placebo added intraoperatively and postoperatively.
- Standard Treatment Group: IV placebo will be initiated during surgery and oral acetaminophen 1000mg every 6 hours will be initiated post-operatively and continued for the duration of the hospital stay (an expected average stay of 2 days) or 48 hours, whichever comes first. Breakthrough pain will be treated with rescue narcotics (IV morphine 2-4mg every 2 hours and oral oxycodone 5-15mg every 4 hours immediately post-operatively through discharge, an expected average stay of 2 days). Hydromorphone (IV 0.5-2 mg every 2 hours and oral 2-4mg every 4 hours) will be used in patients with morphine or oxycodone allergy or intolerance.
  IV placebo: Compare addition of IV placebo intraoperatively and postoperatively against IV Caldolor (ibuprofen) added intraoperatively and postoperatively.
Arm/Group | Opioid-sparing Group | Standard Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/28 | 2/34
Other Adverse Events (participants affected / at risk) | 2/28 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid-sparing Group (N=28) | Standard Treatment Group (N=34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — A disorder characterized by bleeding from the nose.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid-sparing Group (N=28) | Standard Treatment Group (N=34)
hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — elevated level of potassium (K+) in the blood serum. Normal potassium levels are between 3.5 and 5.0 mmol/L (3.5 and 5.0 mEq/L) with levels above 5.5 mmol/L defined as hyperkalemia.
burning at IV site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — I.V. fluid or medications leak into the surrounding tissue.

LIMITATIONS AND CAVEATS:
Groups were not balanced re:patient age, so pain scores were analyzed, including age as a covariate, to account for this difference. A second limitation is that analysis was not powered to detect rare bleeding complications or sellar hematoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT02351700/Prot_SAP_000.pdf